CLINICAL TRIAL: NCT05761028
Title: A Randomized, Double-Blind, Placebo-Controlled Phase Ⅱ/Ⅲ Clinical Study to Evaluate the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Subjects With Moderate to Severe Asthma
Brief Title: A Study of CM310 in Subjects With Moderate to Severe Asthma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-002
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-02

CONDITIONS: Moderate to Severe Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM310 high dose (Experimental): CM310 is injected subcutaneously (SC) with a loading dose at the first dose, and then high dose thereafter, once every 2 weeks (Q2W) for a total of 26 doses.
  Interventions: Drug: CM310
- CM310 low dose (Experimental): CM310 is injected subcutaneously (SC) with a loading dose at the first dose, and then low dose thereafter, once every 2 weeks (Q2W) for a total of 26 doses.
  Interventions: Drug: CM310
- Placebo (Placebo Comparator): Subcutaneous injection (SC), once every 2 weeks (Q2W) for a total of 26 doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CM310 — CM310 Recombinant Humanized Monoclonal Antibody Injection
  Arms: CM310 high dose; CM310 low dose
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled Phase Ⅱ/Ⅲ clinical study to evaluate the efficacy, safety, PK characteristics, PD effects and immunogenicity of CM310 in subjects with moderate to severe asthma.

The study consists of three periods, including an up to 4-week screening period, a 52-week randomized treatment period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the study and voluntarily sign the informed consent form.
2. Age ≥12 and ≤75 years old, male or female, weight ≥40 kg.
3. The subject has been diagnosed with asthma for at least 1 year, and the current disease status meets the diagnostic criteria of GINA 2022.
4. Pre-bronchodilator FEV1 measured ≤ 80% of the normal predicted value at screening and baseline visits (V1 and V2).
5. A positive bronchodilation test (≥12% increase in the FEV1 post-bronchodilator and an absolute FEV1 increase of ≥200 mL) within 24 months before consent or at screening.
6. The subject has received medium-to-high dose ICS combined with at least one control drug, such as LABA, LAMA, LTRA, theophylline, for at least 3 months before signing the informed consent, and maintained stable treatment regimen and dosage for at least 1 month before signing the informed consent.
7. Asthma Control Questionnaire-5 (ACQ-5) score ≥1.5 at screening and baseline visits (V1 and V2).
8. Subjects must have experienced at least one severe asthma exacerbation event within 12 months before consent, and have not experienced a severe asthma exacerbation event within 1 month before consent, with at least one severe asthma exacerbation event occurring during treatment with medium-to-high dose ICS.
9. Subjects (including partners) have no plans to have children and voluntarily use highly effective contraception within 3 months after the last dose of study drug from the date of signing the informed consent.

Exclusion Criteria:

1. Received biological agents with the same therapeutic purpose within 6 months before signing the informed consent.
2. Prior autoimmune disease or inflammatory treatment with biologic agents/systemic immunosuppressive agents within 8 weeks or 5 half- lives (whichever is longer) prior to informed consent.
3. Received immune globulin or blood products within 30 days before informed consent.
4. Subjects treated with systemic corticosteroids (except for topical, ophthalmic, or intranasal corticosteroids) from 4 weeks before signing the informed consent to the date of randomization.
5. Received live or attenuated vaccine within 3 months before informed consent signing or planned to receive live or attenuated vaccine during the study period.
6. Initiation of desensitization therapy within 3 months before informed consent.
7. Underwent bronchial thermoplasty within 12 months before informed consent.
8. Current smokers or former smokers who quit smoking less than 6 months or former smokers who quit smoking more than 6 months with a smoking history of more than 10 pack-years.
9. Chronic obstructive pulmonary disease (COPD) or other lung disease that may impair lung function, as judged by the investigator.
10. Active infection or acute infection requiring systemic anti-infective therapy from 4 weeks before enrollment to the time of randomization.
11. Previous history of known or suspected immunosuppression, including a history of invasive opportunistic infection, even if the infection has resolved; Or the presence of unusual frequent, recurrent, or prolonged infections.
12. History of malignancy: subjects with basal cell carcinoma, localized squamous cell carcinoma of the skin, or carcinoma in situ of the cervix are eligible to enter the study if they have completed curative treatment for at least 12 months before signing the informed consent. Subjects with other malignancies are allowed to enter the study if they have completed curative treatment for at least 5 years before signing the informed consent.
13. The presence of any severe and/or uncontrolled medical condition that in the judgment of the investigator may affect the evaluation of the drug, including but not limited to: severe neurological disease, history of severe mental disorder, major cardiovascular disease, diabetes mellitus poorly controlled by intensive treatment, QTcF interval prolongation, or persistent arrhythmia.
14. Major surgery within 8 weeks prior to informed consent or planned surgery requiring general anesthesia or hospitalization for > 1 day during the study period.
15. Fertile women with positive pregnancy test results during screening; Pregnant or lactating women.
16. Positive screening serologic test for HIV or treponema pallidum.
17. Chronic hepatitis B virus or hepatitis C virus infection.
18. Subjects with abnormal liver and kidney function, such as aspartate aminotransferase or alanine aminotransferase>3 × ULN, or serum creatinine>1.5 × ULN.
19. Have systemic diseases other than asthma that result in an elevated peripheral blood eosinophil count or other diseases such as helminth parasitic infections for which standard treatment is not received or does not respond.
20. Allergy or intolerance to components of CM310 injection or placebo or history of severe drug allergy or anaphylactic shock.
21. Have been enrolled in a clinical trial of any drug or medical device within 3 months before signing informed consent, or are within the follow-up period of a clinical study or the five half-lives of the trial drug (whichever is longer) before signing informed consent.
22. Subjects who have used heavy alcohol within 3 months before screening.
23. History of drug abuse within 5 years before signing informed consent.
24. The investigator considers that there are any conditions that may prevent the subject from completing the study or present a significant risk to the subject or other factors that may reduce the likelihood of enrollment.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2023-04-28 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of severe asthma exacerbations | 52 weeks

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator Forced expiratory volume in 1 second (FEV1) at Week 12 | 56 weeks
Rate of change from baseline in pre-bronchodilator FEV1 at Week 12 | 56 weeks
Change from baseline in FEV1 percentage of predicted value (FEV1% Pred) | 56 weeks
Change from baseline in Peak diurnal and nocturnal expiratory flow (PEF) | 56 weeks
Change from baseline in Forced vital capacity (FVC) | 56 weeks
Change from baseline in Forced Expiratory Flow (FEF) 25-75% | 56 weeks
Change from baseline in FEV1 after the use of bronchodilator | 56 weeks
Annualized rate of subjects experiencing the event of loss of asthma control (LOAC) | 52 weeks
Annualized rate of severe asthma exacerbations leading to hospitalization or emergency department observation | 52 weeks
Time to the first onset of the severe asthma exacerbation event | 52 weeks
Time to the onset of the first event of LOAC | 52 weeks
Change from baseline in the Asthma Control Questionnaire-5 (ACQ-5) score at each evaluation time point | 56 weeks
Change from baseline in asthma symptom score at each evaluation time point | 56 weeks
Change from baseline in the Standardized Asthma Quality of Life Questionnaire (AQLQ(S)) score at each evaluation time point | 56 weeks
Change from baseline in the number of inhalations of SABA | 56 weeks
Incidence of Adverse events (AEs) | 56 weeks
The plasma concentration of CM310 | 56 weeks
Change from baseline in human thymus and activation-regulated chemokine (TARC) | 56 weeks
Change from baseline in total IgE (immunoglobulin E) | 56 weeks
Change from baseline in fractional exhaled nitric oxide (FeNO) | 56 weeks
Anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) | 56 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijin, China

IPD SHARING:
Plan to Share IPD: Undecided